CLINICAL TRIAL: NCT01551186
Title: The Use of the Probiotic, Lactobacillus Rhamnosus GG to Evaluate Colonization With Antimicrobial Resistant Bacteria in High Risk Patients
Brief Title: The Use of Probiotics to Evaluate Colonization With Antimicrobial Resistant Bacteria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201106182; 1U54CK000162 (NIH)
Record Dates: First submitted 2012-03-02; First posted 2012-03-12 (Estimated); Results first posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Infectious Disease of Digestive Tract
Keywords: Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): Patients randomized to probiotic therapy will receive 1 capsule containing 1010 cells of Lactobacillus rhamnosus GG on a twice-daily basis
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG
- Standard of Care (No Intervention): Patients in the control arm will receive standard care

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus GG — 1 capsule containing 10 billion cells of Lactobacillus rhamnosus GG on a twice-daily basis
  Other Names: Culturelle
  Arms: Probiotic

SUMMARY:
The purpose of this study is to evaluate the effectiveness of bacteria called Lactobacillus GG, a Probiotic, in preventing the growth of resistant bacteria in the digestive tract in patients on a ventilator.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old
* Admission to the Medical ICU
* Expected to be on Mechanical Ventilation through an endotracheal tube for >48 hours

Exclusion Criteria:

* Pregnancy
* Immunosuppression
* Prosthetic valve or vascular graft
* Cardiac trauma
* Pancreatitis
* History of rheumatic fever
* Endocarditis or congenital cardiac abnormality
* Gastroesophageal or intestinal injury or foregut surgery during the current admission
* Oropharyngeal mucosal injury
* Placement of a tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria J Fraser, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Kollef MH. Prevention of hospital-associated pneumonia and ventilator-associated pneumonia. Crit Care Med. 2004 Jun;32(6):1396-405. doi: 10.1097/01.ccm.0000128569.09113.fb. PMID 15187525
- [Background] Ruemmele FM, Bier D, Marteau P, Rechkemmer G, Bourdet-Sicard R, Walker WA, Goulet O. Clinical evidence for immunomodulatory effects of probiotic bacteria. J Pediatr Gastroenterol Nutr. 2009 Feb;48(2):126-41. doi: 10.1097/MPG.0b013e31817d80ca. PMID 19179874
- [Background] de Smet AM, Hopmans TE, Minderhoud AL, Blok HE, Gossink-Franssen A, Bernards AT, Bonten MJ. Decontamination of the digestive tract and oropharynx: hospital acquired infections after discharge from the intensive care unit. Intensive Care Med. 2009 Sep;35(9):1609-13. doi: 10.1007/s00134-009-1554-9. Epub 2009 Jun 24. PMID 19551370
- [Background] Oostdijk EA, de Smet AM, Blok HE, Thieme Groen ES, van Asselt GJ, Benus RF, Bernards SA, Frenay IH, Jansz AR, de Jongh BM, Kaan JA, Leverstein-van Hall MA, Mascini EM, Pauw W, Sturm PD, Thijsen SF, Kluytmans JA, Bonten MJ. Ecological effects of selective decontamination on resistant gram-negative bacterial colonization. Am J Respir Crit Care Med. 2010 Mar 1;181(5):452-7. doi: 10.1164/rccm.200908-1210OC. Epub 2009 Dec 3. PMID 19965807

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Probiotic | Standard of Care
Started | 50 | 53
Completed | 30 | 40
Not Completed | 20 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotic | Standard of Care | Total
Number analyzed (Participants) | 30 | 40 | 70
Age, Continuous [Median (Full Range); unit: years] | 65 [29 to 82] | 59 [32 to 82] | 60 [29 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 12 | 20 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White race | 19 | 24 | 43
  Race: Non-white race | 11 | 16 | 27
Region of Enrollment [Number; unit: participants]
  United States | 30 | 40 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Combination of Gastrointestinal Tract Colonization With Multi-drug Resistant Gram-negative Bacteria, C. Difficile and VRE
Description: Colonization of the gastrointestinal tract with C. difficile, vancomycin-resistant enterococci, multidrug-resistant Acinetobacter baumannii, and multidrug- resistant Pseudomonas. Colonization occurs when the subject acquires the above organism while in the study.
Time Frame: Participants will be followed while Intubated, an expected average of 7 days. The outcome will be measured 3 days after enrollment and at the end of intubation, average time 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic | Standard of Care
Number analyzed (Participants) | 30 | 40
Participants | 8 | 8

ADVERSE EVENTS:
Arm/Group | Probiotic | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/40
Other Adverse Events (participants affected / at risk) | 0/30 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No